CLINICAL TRIAL: NCT03835689
Title: Parent Training for Challenging Behaviour in Children with Neurodevelopmental Disabilities: Strongest FamiliesTM Neurodevelopmental
Brief Title: Strongest FamiliesTM Neurodevelopmental
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McGill University (Other); University of Alberta (Other); Child-Bright Network (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB#1023970
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2022-03

CONDITIONS: Neurodevelopmental Disorders; Behavior Disorders
Keywords: Behavioural intervention; E-health intervention; Parenting intervention
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician conducting analysis will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Strongest Families Program Self-Managed (no coaching) (Experimental): They will receive Strongest Families intervention immediately as well as the usual care services available for the 10 month study period.
  Interventions: Behavioral: Strongest Families Intervention (formerly Family Help)
- Strongest Families Program with Group Telephone Coaching (Experimental): They will receive Strongest Families intervention immediately as well as the usual care services available for the 10 month study period.
  Interventions: Behavioral: Strongest Families Intervention (formerly Family Help)
- Information Resource Website (No Intervention): They will not receive Strongest Families Intervention during the 10 month study phase, but will receive the usual care services and access to an Information Resource Website.

INTERVENTIONS:
Behavioral: Strongest Families Intervention (formerly Family Help) — Distance HEALTH education intervention focused on skill learning for parents
  Other Names: Formerly the Family Help Program
  Arms: Strongest Families Program Self-Managed (no coaching); Strongest Families Program with Group Telephone Coaching

SUMMARY:
Children and adolescents with neurodevelopmental conditions are 3 to 5 times more likely than their peers to have other mental disorders such as anxiety, depression and disruptive behaviour. Furthermore, these conditions are less likely to be recognized, diagnosed and treated than for typically developing children. Parent training is a well-established approach to help parents change their behaviour and communication with their children with the goal of improving child behaviours. Parent-focused programs that are designed for typically developing children have shown mixed results for children with neurodevelopmental conditions and parents have reported significant challenges in accessing traditional health services due to barriers to care. There is an urgent need to explore how effective distance-delivered parenting programs can be implemented in real-world settings and how they should be adapted to meet the needs of families with children with neurodevelopmental conditions. The goal of this research project is to develop and test the effectiveness of two versions (group coaching & self-managed) of an online parenting program for managing challenging behaviours in children with neurodevelopmental disabilities. The Strongest Families Neurodevelopmental program is based on the well-established Strongest Families Parenting program for typically developing children with challenging behaviours, adapted with substantial involvement from a pan-Canadian Parent Advisory Committee. The program consists of 11 skill-based sessions with demonstration videos, audio clips, exercises, a resource webpage and a Parent-to-Parent online group (a closed Facebook group).

ELIGIBILITY:
SCREENING: Parents/caregivers must meet all of the following criteria to be eligible to proceed to Consent:

1. Have a child between 3-14 years of age with a diagnosis of a neurodevelopmental disorder (i.e. Autism Spectrum Disorder, Cerebral Palsy, Epilepsy, Global Developmental Delay, Down Syndrome, Fetal Alcohol Spectrum Disorder (FASD), severe learning disability or any other diagnosis that influences how their child gets around, communicates their ideas, processes what they hear, or remembers things as reported by parents/caregivers).
2. The child has been experiencing behavioural problems that interfere with the activities of daily living (as defined by the caregiver) for at least 6 months prior to study screening.
3. Have been the primary caregiver for a minimum of 6 months prior to entry into the study.
4. Have a reasonable expectation of being be the primary caregiver for at least 10 months after study enrolment.
5. Read, write, and understand English.
6. Have access to a telephone.
7. Have regular access to a tablet, smartphone or computer connected to high speed Internet.
8. Live in Canada.
9. Commit to the requirements of taking part in the study (e.g. available to attend weekly coaching calls, having a Facebook account to access Parent-to-Parent support group)

Any of the following criteria will exclude individuals from proceeding to Consent:

1. Child is NOT able to understand everyday language and instructions or communicate needs as reported by parent/caregiver.
2. Parent or child has ongoing struggles with symptoms of psychosis, schizophrenia, bipolar disorder or major depression (i.e. the symptoms are not well managed).
3. Child is at imminent risk of serious harm to self or others (i.e. requiring hospitalization or medical attention).
4. Child regularly engages in moderate to severe self-injurious behaviours, as reported by the parent.
5. Child has attempted suicide in the past 6 months.
6. Parent has previously taken part in a Strongest Families Parenting Program.
7. Parent has taken part in Triple P, COPE, Incredible Years or another parent training program within 6 months prior to starting the study.

BASELINE ASSESSMENT:

1. Meet minimum score of 16 (for ages 2 - 4 years) or 17 (for ages 4-17) on the Total Difficulties Score of the Strengths and Difficulties Questionnaire.
2. Meet a minimum level of child's cognitive functioning as determined by the question* below. Parents must endorse 1, 2 or 3 on the following question:

Compared with children of the same age, does your child have difficulty learning things? Would you say your child has: no difficulty, some difficulty, a lot of difficulty or cannot do at all? No difficulty........................ 1 Some difficulty....................2 A lot of difficulty..................3 Cannot do at .....................4

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline parenting self-efficacy at 5 month post-randomization | Baseline and 5 month post-randomization
  Statistically significant improvement in parent report of self-efficacy from baseline to 5 month follow up for both intervention groups compared to control, as measured by the total score on the Self-Efficacy subscale of the Child Adjustment and Parent Efficacy Scale - Developmental Disability (CAPES-DD) questionnaire. The CAPES-DD assesses emotional and behavioural problems in children with developmental disabilities (age 2 - 16 years) and their parents' self-efficacy to manage specific problematic behaviours. For each of 16 problem child behaviours, respondents are asked to rate their confidence in their ability to successfully manage the behaviour. Ratings range on a scale from 1 ('certain I can't manage it') to 10 ('certain I can manage it'). Total scores range from 16 - 160 with higher scores indicating greater levels of parent self-efficacy.
Change from baseline child's emotion regulation at 5 month post-randomization | Baseline and 5 month post-randomization
  Statistically significant improvement in emotion regulation from baseline to 5 months for both intervention groups compared to control, as measured by the total score of the Emotion Regulation Checklist (ERC). The 24-item scale consists of two subscales: Lability/Negativity characterized by inflexibility, mood swings and dysregulated negative affect (e.g., "is prone to angry outbursts/tantrums easily"), and Emotion Regulation representing appropriate affect, empathy and awareness of one's emotions (e.g., "responds positively to neutral or friendly approaches by peers'). Parents are asked to report, on a 4 point Likert-type scale ranging from Never to Almost Always, how much each statement applies to their child. An overall emotional regulation score is calculated by reverse scoring the Emotion Regulation items and summing all questionnaire items; a higher score indicating more dysregulation. We will use total scores which range from 23 - 92 (item 12 is not used in the calculation).

SECONDARY OUTCOMES:
Change from baseline parenting self-efficacy at 10 month post-randomization | Baseline and 10 month post-randomization
  Statistically significant improvement in parent report of self-efficacy from baseline to 10 month follow up for both intervention groups compared to control, as measured by the total score of the Self-Efficacy subscale of the Child Adjustment and Parent Efficacy Scale - Developmental Disability (CAPES-DD) questionnaire. The CAPES-DD assesses emotional and behavioural problems in children with developmental disabilities (age 2 - 16 years) and their parents' self-efficacy to manage specific problematic behaviours. For each of 16 problem child behaviours, respondents are asked to rate their confidence in their ability to successfully manage the behaviour. Ratings range on a scale from 1 ('certain I can't manage it') to 10 ('certain I can manage it'). Total scores range from 16 - 160 with higher scores indicating greater levels of parent self-efficacy.
Change from baseline child's emotion regulation at 10 month post-randomization | Baseline and 10 month post-randomization
  Statistically significant improvement in emotion regulation from baseline to 10 months for both intervention groups compared to control, as measured by the total score of the Emotion Regulation Checklist (ERC).The 24-item scale consists of two subscales: Lability/Negativity characterized by inflexibility, mood swings and dysregulated negative affect (e.g., "is prone to angry outbursts/tantrums easily"), and Emotion Regulation representing appropriate affect, empathy and awareness of one's emotions (e.g., "responds positively to neutral or friendly approaches by peers'). Parents are asked to report, on a 4 point Likert-type scale ranging from Never to Almost Always, how much each statement applies to their child. An overall emotional regulation score is calculated by reverse scoring the Emotion Regulation items and summing all questionnaire items; a higher score indicating more dysregulation. We will use total scores which range from 23 - 92 (item 12 is not used in the calculation).
Reduced children's externalizing behaviours | Baseline, 5 and 10 month post-randomization
  Statistically significant reduction in child's behavior problems between baseline and 5 months and baseline and 10 months for both interventions groups compared to control, as measured by the Difficulties score of the Strengths and Difficulties Questionnaire (SDQ). The SDQ measures children's emotional problems, conduct disorder, hyperactivity, peer problems and prosocial behavior. The Total Difficulties scores is calculated by summing all scores except items on the prosocial scale. Scores range from 0 - 40 with higher scores indicating more problematic behavior.
Improved parental well-being | Baseline, 5 and 10 month post-randomization
  Statistically significant reduction of parent report of depression, anxiety and stress from baseline to 5 months and baseline to 10 months for both interventions groups compared to control, as measured by total score of the Depression, Anxiety, Stress Scale - 21 (DASS-21). The DASS-21 measures severity of symptoms related to depression, anxiety and stress. Respondents rate how much each symptom applied to them in the past week using a scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Total scores are calculated by summing responses and multiplying by 2 to allow comparison to severity scores established with the long form of the DASS which has 42 items (e.g. normal to extremely severe). Scores range from 0 - 126, with higher scores indicating more distress.
Incremental Cost-Effectiveness Ratio (ICER) - Child | Baseline, 5 and 10 month post-randomization
  ICER are calculated by dividing the difference in cost by the difference in effectiveness when comparing two interventions and represent the additional cost or savings associated with gaining or losing an additional unit of effectiveness. To assess the value for money of an intervention relative to another, decision-makers can compare ICER values to the amount their jurisdiction would be willing to pay to gain or willing to accept to forgo a unit of the effectiveness outcome that was included in the ICER. Cost will be measured in Canadian dollars and effectiveness will be measured using quality adjusted life years (QALY). Cost and effectiveness will reflect those of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD, Principal Investigator — IWK Health Centre; Lucyna Lach, PhD, Principal Investigator — McGill University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to indicate during Informed Consent whether their de-identified data may be shared with other researchers, provided the study is approved by an ethics board and researchers agree to use the data only for the purposes described in the approved research study. De-identified data from all outcome measures will be made available to approved researchers upon request, provided individual participants have provided consent.
Supporting Information: Study Protocol, SAP, ICF